CLINICAL TRIAL: NCT05033548
Title: Technology Enabled And Molecular Monitoring of the Allograft and Transplant rEcipient
Acronym: TEAMMATE
Status: Terminated | Type: Observational
Why Stopped: Decision by Sponsor after careful review of study data available.
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00018
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-06

CONDITIONS: Transplant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Managed with AlloCare Monitoring
- Managed with Standard of Care

SUMMARY:
The primary objective of the study is to assess the impact of AlloCare mHealth remote monitoring on the early post-transplant period in solid organ transplantation.The outcome measure for primary objective is overall reduction in Readmission Rate to hospital in 90 days for all causes. Patients will be assessed across 4 different organ groups (Kidney, Liver, Lung and Heart Transplantation). The secondary objective is to consider the impact of mHealth and app-based monitoring on variables known to impact long term outcomes over the first 12 months post transplantation, as well as impact on quality of life. The outcome measures for secondary objective are: 1. Tacrolimus Variability (Time in Therapeutic Range,) as a surrogate to adherence and compliance 2. BPAR within 3,6, and 12 months 3. Patient satisfaction at 90 days 4. SF-36 change at 90 days 5. HbA1c monitoring (diabetic patients only)

DETAILED DESCRIPTION:
If a patient is randomized to the AlloCare App arm and does not have access to a smartphone to utilize AlloCare App, a device will be provided for the duration of the study for use, with the AlloCare app installed. Otherwise, patients will be allowed to use their own device . The device and data plan will be covered by the sponsor for the duration of the study. Enrollment on the Allocare app with weekly transmission of patient data to the transplant programs is expected. In addition, all patients will have AlloSure dd-cfDNA surveillance per their institutional schedule. These patients will be compared to the current standard: Paper binder, with written diary, also including AlloSure with weekly visits as needed per center protocol.

Patients will follow an AlloSure cfDNA testing schedule based on medical necessity and outlined as the standard of care by the institution. The mHealth remote monitoring is weekly for the first 90 days and then monthly until 12 months post-transplant. The remainder of the schedule will follow the current standard of care.

If study sites are unable to follow this recommend schedule, please create an amended schedule of events for review by the sponsor. DSA (optional) is aimed to be collected as part of their post-transplant surveillance. The EMR will be examined at 3,6, and 12 months post transplantation.

The AlloCare App is a smart phone-based app that empowers transplant patients to manage their health by enabling them to adhere to and track their health activities and transmit data on their compliance to their care team & community providers. Primary functionality of the application involves medication management, which includes up to date medication lists derived directly from the EHR, scheduling of medication and medication reminders and adherence tracking. In addition, the user can record and monitor other wellness activities such as water intake, steps, mood, sleep etc. Support for testing adherence is provided by allowing the user to connect to patient care managers directly through the app, schedule both in-center and mobile blood-draws and providing lab visit reminders. Lastly, the app provides the user with support through multi-modality educational materials and a virtual connection to a community of other post-transplant patients, as well as to their own care givers.

Patients will also be offered mobile phlebotomy if they are unable to visit a local lab. This is a service provided by CareDx for all patients needing Allosure test for clinical decision making. The mobile blood draw will be ordered by your providers as clinically necessary and coordinated by CareDx, which will draw all regular tests, urine sample as well as the AlloSure. Results are couriered to your lab of choice for analysis. This can be your own hospital lab so you can directly see the results in your hospital EMR. AlloSure results will be sent to the center in the same format as you are currently receiving them. Patients utilizing AlloCare App for post-transplant monitoring will be able to review their Allosure results on the App.

For investigators who do not have an electronic medical record (EMR) with transplant functionality and/or a fully functional transplant management database, the OTTR SaaS platform is an option that can be provided for the duration of the investigation, to allow capture of all critical data fields. OTTR SaaS is a fully HIPAA compliant Transplant patient management application with pre- and post-transplant longitudinal workflow management and data capture capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 12 years or above. (Gillick Competent)

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

* Participant who is pregnant, lactating or planning pregnancy during the trial.
* Significant hepatic impairment (determined by the PI)
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Participant with life expectancy of less than 6 months, or inappropriate for diagnostic monitoring through regular blood sampling.
* >3 months post-transplant
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational pharmaceutical product in the past 12 weeks.
* Multi-organ transplant (e.g., Kidney-Pancreas).
* Recipients of a transplant from a monozygotic (identical) twin
* Recipient of non-autologous bone marrow transplant
* Patients with a history of needle phobia.
* Patients who are not English or Spanish speaking

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a single solid organ transplant of either Lung, Liver, Kidney or Heart, will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Overall reduction in Readmission Rate to hospital within 90 days (all causes) | 90 days
  The aim of this study is to evaluate AlloCare and remote patient monitoring developed as an integrated mHealth service, assessing whether the combination of app and monitoring deployed within the solid organ transplant population can help support durable behavioral changes in patients that improve self-care and shared decision-making within the patient-provider relationship.

SECONDARY OUTCOMES:
Tacrolimus Variability (Time in Therapeutic Range,) at 3,6, and 12 months as a surrogate to adherence and compliance | 3, 6, and 12 months
  Use of Allocare is hoped to empower patient self-care with improved monitoring with result in fewer readmissions after transplant and reduced clinic visits, better medication adherence, and fewer immunosuppression related complications when compared to standard of care.
BPAR at 3, 6, and 12 months | 3, 6, and 12 months
  Use of Allocare is hoped to empower patient self-care with improved monitoring with result in fewer readmissions after transplant and reduced clinic visits, better medication adherence, and fewer immunosuppression related complications when compared to standard of care.
Patient satisfaction at 90 days | 90 days
  Use of Allocare is hoped to empower patient self-care with improved monitoring with result in fewer readmissions after transplant and reduced clinic visits, better medication adherence, and fewer immunosuppression related complications when compared to standard of care. In addition, use of the app will lead to improved patient and provider satisfaction at 90 days.
SF-36 change at 90 days | 90 days
  Use of Allocare is hoped to empower patient self-care with improved monitoring with result in fewer readmissions after transplant and reduced clinic visits, better medication adherence, and fewer immunosuppression related complications when compared to standard of care.
HbA1c monitoring (diabetic patients only) at 3,6, and 12 months | 3, 6, and 12 months
  Use of Allocare is hoped to empower patient self-care with improved monitoring with result in fewer readmissions after transplant and reduced clinic visits, better medication adherence, and fewer immunosuppression related complications when compared to standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Shimul Shah, M.D., Principal Investigator — University of Cincinnati
Locations (10):
- United States (10):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - ECMC State University of NY/University of Buffalo, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin